CLINICAL TRIAL: NCT03450187
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Multiple Ascending-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral TP-271 in Healthy Adult Subjects
Brief Title: A Phase 1 TP-271 Oral PK Multiple Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TP-271-004
Record Dates: First submitted 2018-02-16; First posted 2018-03-01 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — TP-271

STUDY DESIGN:
Intervention Model Description: Up to 5 cohorts of 8 subjects each will be enrolled. Subjects in each cohort will be randomized 6:2 to receive multiple oral doses of TP 271 at 1 of 5 ascending doses of TP-271 or placebo once or twice daily for 7 days, as shown in the table below. Every effort will be made to dose all subjects in a cohort on the same day.
  Proposed Oral Doses of Study Drug by Dose Cohort Cohort Dose Regimen Proposed Oral Dose A Once daily 50 mg TP-271 q24 (n = 6) or matching placebo (n = 2) B Once daily 100 mg TP-271 q24 (n = 6) or matching placebo (n = 2) C Once daily 200 mg TP-271 q24 (n = 6) or matching placebo (n = 2) D Once daily 300 mg TP-271 q24 (n = 6) or matching placebo (n = 2) E Once daily 400 mg TP-271 q24 (n = 6) or matching placebo (n = 2) Abbreviations: q24 = every 24 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A (Active Comparator): 50 mg TP-271 q24 (n=6), a novel, broad-spectrum tetracycline-class antibiotic or matching placebo (n=2) once daily for 7 days.
  Interventions: Drug: TP-271
- Cohort B (Active Comparator): 100 mg TLP-271 q24 (n=6), a novel, broad spectrum tetracycline-class antibiotic or matching placebo (n=2) once daily for 7 days.
  Interventions: Drug: TP-271
- Cohort C (Active Comparator): 200 mg TP-271 q24 (n=6), a novel, broad spectrum tetracycline-class antibiotic or matching placebo (n=2) once daily for 7 days.
  Interventions: Drug: TP-271
- Cohort D (Active Comparator): 300 mg TP-271 q24 (n=6), a novel, broad spectrum tetracycline-class antibiotic or matching placebo (n=2) once daily for 7 days.
  Interventions: Drug: TP-271
- Cohort E (Active Comparator): 400 mg TP-271 q24 (n=6), a novel, broad spectrum tetracycline-class antibiotic or matching placebo (n=2) once daily for 7 days.
  Interventions: Drug: TP-271

INTERVENTIONS:
Drug: TP-271 — multiple oral doses of TP-271 or placebo, randomized 6:2, doses escalating 50 mg, 100 mg, 200 mg, 300 mg, 400 mg once daily for 7 days.

SUMMARY:
This is a phase 1, single-center, randomized, placebo-controlled, double-blind, multiple ascending-dose study to assess the safety, tolerability, and PK of oral TP-271 in healthy adult subjects. Male or female subjects aged 18 to 50 years who fulfill the inclusion/exclusion criteria will be enrolled in this study.

DETAILED DESCRIPTION:
This is a phase 1, single-center, randomized, placebo-controlled, double-blind, multiple ascending-dose study to assess the safety, tolerability, and PK of oral TP-271 in healthy adult subjects. Male or female subjects aged 18 to 50 years who fulfill the inclusion/exclusion criteria will be enrolled in this study.

Up to 5 cohorts of 8 subjects each (up to a total of 40 subjects) will be enrolled. Subjects in each cohort will be randomized 6:2 to receive multiple oral doses of TP 271 or placebo. Every effort will be made to dose all subjects in a cohort on the same day.

Doses of study drug will be administered orally either once daily in the morning or twice daily in the morning and evening from Days 1 to 7. In all subjects, the morning dose will be administered following an overnight fast (minimum 8 hours) of food and all beverages, except for water. For subjects in Cohorts D and E only, the evening dose will be administered following a minimum 3-hour fast of food and all beverages, except for water. Fasting in all cohorts will continue for at least 2 hours following each study drug administration.

During the Screening Period (within 28 days prior to the subject receiving study drug), each subject will be assessed for eligibility. Each subject must sign and date an ICF prior to undergoing any study-related procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Be within the age range of 18 to 50 years, inclusive, at the time of Screening
2. Voluntarily sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved ICF to participate in the study after all relevant aspects of the study have been explained to and discussed with the subject and before undergoing any study-related procedures
3. Have a body mass index (BMI) ≥18.0 and ≤33.0 kg/m2
4. Have a negative history of and negative screening results for human immunodeficiency virus (HIV) types 1 and 2 and hepatitis B and C
5. Have the ability to communicate with the study unit staff in a manner sufficient to carry out all protocol procedures as described
6. Female subjects must be of non-childbearing potential, either 1-year postmenopausal or surgically sterile (i.e., bilateral oophorectomy, bilateral tubal ligation, or complete hysterectomy)
7. Male subjects must be willing and able to use a barrier method of contraception or practice abstinence (including male subjects who had a vasectomy) from dosing to 90 days after final administration of the study drug

Exclusion Criteria:

1. History and/or presence of any clinically significant disease or disorder, such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal, endocrine, psychiatric or mental disease or disorder, or mental or legal incapacitation, which, in the opinion of the PI, may either put the subject at risk due to participation in the study, influence the results of the study, or influence the subject's ability to participate in the study
2. Clinical laboratory values that fall outside of the eligibility range specified in Appendix D are exclusionary; for clinical laboratory values that are not included in Appendix D, values outside of the reference range are exclusionary, except for those parameters listed in Table 4).

   Table 4 Acceptable Out-of-Range Clinical Laboratory Values

   Low Chemistry Values:

   Bicarbonate (a) Chloride GGT HDL cholesterol LDH LDL cholesterol Phosphorus

   High Chemistry Values:

   Chloride HDL cholesterol LDL cholesterol Phosphorus Triglycerides

   Out-of-Range Urinalysis Values; High or low specific gravity Cloudy Mucus Crystals Ketones (b) Hyaline casts High or low pH Urobilinogen (c)

   Out of Range Hematology Values; High hematocrit Basophils Monocytes MCV MCH MCHC RBC

   a Bicarbonate >18 mEq/L. b Acceptable only when the concurrent blood glucose is normal. c Measured when monitoring the serum bilirubin concentration. Abbreviations: GGT = gamma-glutamyltransferase; HDL = high-density lipoprotein; LDH = lactate dehydrogenase; LDL = low-density lipoprotein; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = mean corpuscular volume; RBC = red blood cell.
3. Known allergy to tetracycline antibiotics or any of the excipients in TP 271
4. Clinically significant abnormality on a 12-lead ECG, which includes the following:

   * Rhythm other than sinus
   * Corrected QT interval using Fridericia's formula (QTcF) >450 msec
   * Evidence of second- or third-degree atrioventricular (AV) block
   * Pathological Q-waves (defined as a Q-wave >40 msec or depth >0.4 to 0.5 mV)
   * Evidence of ventricular pre-excitation
   * Evidence of complete left bundle branch block (BBB), right BBB, or incomplete left BBB
   * Intraventricular conduction delay with QRS duration >120 msec
   * ST segment abnormalities, unless judged by the PI to be nonpathologic
5. History of seizures
6. History within 3 years of a positive result on a urine screen for drugs of abuse or a positive result on a urine screen at Screening for any of the following drugs of abuse: tetrahydrocannabinols, cocaine, opioids, phencyclidines, amphetamines, benzodiazepines, barbiturates, and cotinine
7. Use of tobacco, nicotine, or nicotine-replacement products within 3 months prior to initial administration of study drug to the EOS Visit
8. Typical weekly alcohol consumption of 7 or more alcoholic drinks, where 1 alcoholic drink is defined as 1 glass of beer (approximately 10 to 12 oz), 1 can of beer (12 oz), 1 glass of wine (approximately 4 to 5 oz), or distilled spirits (approximately 1 oz or 30 mL of liquor)
9. Alcohol consumption within 48 hours prior to admission
10. Participation in a clinical study within 10 half-lives of the prior study treatment or within the previous 3 months (if the half-life of investigational agent is unknown) prior to initial administration of study drug or planned participation in another clinical study concurrent with the present study
11. History of difficulty donating blood or poor venous access
12. Recent blood donation (1 unit or approximately 525 mL) within 1 month prior to receiving study drug or plans to donate prior to receiving study drug or during the clinical study
13. Use of any prescription or nonprescription medication, including vitamins or herbal medications, vaccination, or immunization within 7 days or 5 half-lives (if known), whichever is longer, prior to initial administration of study drug, with the following exceptions: medications used to treat an AE are permitted, and the use of acetaminophen, naproxen, and ibuprofen is permitted, except for within 24 hours prior to dosing
14. Male subjects who donate or plan to donate sperm during the study or within 90 days after final administration of the study drug
15. Unwillingness or inability to follow the procedures outlined in the clinical study protocol
16. Previous participation in another TP-271 study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From the time of signing of the informed consent form throughout study completion (approximately 39 days)
  Incidence, intensity, and type of adverse events.
A Directed Physical Examination including chest/respiratory | Day -1 to the End of Study visit, Day 21
  changes in physical examination findings for chest/respiratory
A Directed Physical Examination including heart/cardiovascular | Day -1 to the End of study visit, Day 21
  Changes in Physical Examination including heart/cardiovascular
Vital Signs including Pulse Rate | Day -1 to the End of study visit, Day 21
  Changes in Pulse Rate
Vital Signs including respiration rate | Day -1 to the End of study visit, Day 21
  Changes in respiration rate
Vital Signs including body temperature | Day -1 to the end of study visit, Day 21
  Changes in body temperature
Vital Signs including blood pressure | Day -1 to the End of study visit, Day 21
  Changes in blood pressure
ECG measurements including PR interval | Day -1 to the End of study visit, Day 21
  Changes in PR interval > or=20
ECG measurements including QRS interval | Day -1 to the end of study visit, Day 21
  Changes in QRS interval> or=10
ECG measurements including QTcF interval | Day -1 to the end of study visit, Day 21
  Changes in QTcF interval 30 to 60, > or =60
Safety Laboratory results including clinical chemistry | Day -1 to the End of study visit, Day 21
  Changes in safety laboratory results including clinical chemistry
Safety Laboratory results including electrolytes | Day -1 to the End of study visit, Day 21
  Changes in safety laboratory results including electrolytes
Safety Laboratory results including hematology | Day -1 to the End of study visit, Day 21
  Changes in safety laboratory results including hematology
Safety Laboratory results including blood glucose | Day -1 to the End of study visit, Day 21
  Changes in Safety laboratory results including glucose
Safety Laboratory results including coagulation | Day -1 to the End of study visit, Day 21
  Changes in Safety Laboratory results including coagulation

SECONDARY OUTCOMES:
Plasma concentrations | Days 1-7
  Plasma concentrations of TP-271 and its C-4 epimer TP-9555 for PK analysis
Urine pharmacokinetics | Days 1-7
  Urine concentrations of TP-271 and it's C-4 epimer, TP-9555
PK parameters - Cmax | Days 1-7
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Cmax (the maximum observed plasma concentration)
PK parameters- Tmax | Days 1-7
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Tmax
PK parameters AUC (0-last) | Days 1-7
  Area under the concentration versus time curve (AUC) from time zero to the last measured time point
PK parameters - AUC (0-inf) | Days 1-7
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC (0-inf) (The area under the concentration vs time curve from time zero extrapolated to infinity)
PK parameters- AUC% extrapolated | Days 1-7
  PL parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC% extrapolated (the percentage of AUC 90-inf) accounted for by extrapolation)
PK parameters - AUC (0-24) | Days 1-7
  AUC from time zero to 24 hours (AUC 0-24)
PK parameters - Lambda-z | Days 1-7
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Lambda-z (Slope of the regression line passing through the apparent elimination phase in a concentration vs time plot)
PK parameters - CL | Days 1-7
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for CL (Clearance: the volume of plasma cleared per unit time)
PK parameters - Vd | Days 1-7
  PK parameters will be calculated using the apparent volume of distribution following oral dosing
PK parameters -T 1/2el | Days 1-7
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for T1/2el (The elimination half-life)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Tsai, MD, Study Director — Tetraphase Pharmaceuticals
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided